CLINICAL TRIAL: NCT04123873
Title: Effect of Combinations of Paracetamol, Ibuprofen, and Dexamethasone on Patient-Controlled Morphine Consumption in the First 24 Hours After Total Hip Arthroplasty. The RECIPE Randomized Clinical Trial
Brief Title: Effect of Combinations of Paracetamol, Ibuprofen, and Dexamethasone on Patient-Controlled Morphine Consumption in the First 24 Hours After Total Hip Arthroplasty
Acronym: RECIPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-JOAST-2019
Record Dates: First submitted 2019-09-27; First posted 2019-10-11 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Hip Arthropathy; Analgesia; Postoperative Pain
Keywords: RECIPE; Hip arthroplasty; Postoperative pain; Analgesia; Multimodal analgesia; Non-opioid analgesia; Acute pain
MeSH Terms: conditions — Acute Pain; Agnosia; Pain, Postoperative | interventions — Acetaminophen; Ibuprofen; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medication will be masked by the pharmacy. The experimental medicine will be packed and labelled by Skanderborg Pharmacy in accordance with the Good Manufacturing Practice regulations. The sponsor has a set of sealed, opaque envelopes with the participants' allocation, and these will only be revealed for the investigators when the data has been analysed and abstracts and conclusions covering the different possibilities for interpreting the trial results, have been agreed upon by the steering committee
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Paracetamol 1000 mg + Ibuprofen 400 mg administered orally 1 hour before surgery and given with 6-hour intervals to a total of 4 times the first postoperative day.
  Plus placebo (matching DXM) IV administered after induction of anaesthesia
  Interventions: Drug: Paracetamol; Drug: Ibuprofen; Drug: Placebo IV
- Group B (Experimental): Paracetamol 1000 mg and placebo (matching ibuprofen) orally 1 hour before surgery and given with 6-hour intervals to a total of 4 times the first postoperative day.
  Plus DXM 24 mg IV after induction of anaesthesia
  Interventions: Drug: Paracetamol; Drug: Dexamethasone; Drug: Placebo oral capsules
- Group C (Experimental): Placebo (matching paracetamol) + ibuprofen 400 mg orally 1 hour before surgery and given with 6-hour intervals to a total of 4 times the first postoperative day.
  Plus DXM 24 mg IV after induction of anaesthesia
  Interventions: Drug: Ibuprofen; Drug: Dexamethasone; Drug: Placebo oral capsules
- Group D (Experimental): Paracetamol 1000 mg + ibuprofen 400 mg orally 1 hour before surgery and given with 6-hour intervals to a total of 4 times the first postoperative day.
  Plus DXM 24 mg IV after induction of anaesthesia
  Interventions: Drug: Paracetamol; Drug: Ibuprofen; Drug: Dexamethasone

INTERVENTIONS:
Drug: Paracetamol — 1g x 4 p.o.
  Other Names: Acetaminophen
  Arms: Group A; Group B; Group D
Drug: Ibuprofen — 400mg x 4 p.o.
  Arms: Group A; Group C; Group D
Drug: Dexamethasone — 24mg IV x 1 after induction om anaesthesia
  Arms: Group B; Group C; Group D
Drug: Placebo oral capsules — p.o. x 4
  Arms: Group B; Group C
Drug: Placebo IV — IV x 1
  Arms: Group A

SUMMARY:
Multimodal pain management is essential for recovery after surgery, aiming to target different pain mechanisms to minimize opioid usage and opioid-related adverse effects. Evidence for benefits and harms of various non-opioid analgesic combinations is, however, nearly non-existing, and large-scale trials are urgently needed.

Recently, the investigators have demonstrated that combining paracetamol and ibuprofen is superior to each single drug when assessing pain after hip replacement. Further improvement is needed, investigating additional non-opioid analgesics to this combination. Glucocorticoids have anti-emetic and analgesic properties, but evidence for analgesic efficacy in combination with paracetamol and ibuprofen is lacking.

The RECIPE trial is an investigator-initiated randomized, placebo-controlled, parallel, 4-group, blinded multicentre trial with 90-day follow-up investigating benefits and harms of different combinations of paracetamol, ibuprofen, and dexamethasone for patients undergoing total hip arthroplasty.

The primary outcome is total use of IV morphine 0-24 hours postoperatively. Secondary outcomes are pain (upon mobilisation, at rest, and during 5 m walk), and adverse events. Exploratory outcomes include quality of sleep, opioid-related adverse effects, serious adverse events (< 90 days), and patient reported disability score and quality of life (at 90 days).

Based on sample-size calculations, 1060 patients are needed to detect a minimal clinically important difference in 24-hour morphine consumption of 8 mg, using a familywise type 1 error rate of 0.05 and a type 2 error rate of 0.2. The primary analyses will be based on the intention to treat population. More than six Danish university- and regional hospitals will participate in the trial.

With this trial the investigators expect to lay the foundation for the best postoperative multimodal analgesic regimen for both total hip arthroplasty and possibly other surgeries, thereby facilitating recovery for millions of future surgical patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective, unilateral, primary THA
* Age ≥ 18
* ASA 1-3
* BMI > 18 and < 40
* Negative urine HCG pregnancy test and use of anti-conception for women in the fertile age
* Give written informed consent to participate in the trial after having fully understood the contents of the protocol and restrictions

Exclusion Criteria:

* Patients who cannot cooperate with the trial
* Concomitant participation in another trial involving medication
* Patients who cannot understand or speak Danish
* Patients with allergy to medication used in the trial
* Patients with daily use of high dose opioid (> oral morphine 30 mg/day or oxycodone 30 mg/day or tramadol 150 mg/day) or any use of other opioids including methadone and transdermal opioids.
* Patients with daily use of systemic glucocorticoids (within 3 months before the trial)
* Contraindications against ibuprofen or paracetamol, for example previous ulcer, known heart failure, known liver failure, or known renal failure (eGRF < 60 ml/kg/1,73m2), known thrombocytopenia (< 100 x 109/l); or against treatment with glucocorticoids
* Dysregulated diabetes (investigator's judgement)
* Patients suffering from alcohol and/or drug abuse - based on the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | 0-24 hours after end of surgery
  Cumulative opioid consumption in units of intravenous morphine equivalents in the first 24 postoperative hours. This includes opioids administered as (a) patient-controlled analgesia (PCA); (b) supplemental opioid administered at the post-anaesthesia care unit the first hour after end of surgery (general anaesthesia) or the first hour after ceasing of spinal anaesthesia; and (c) any supplemental opioid given at the ward

SECONDARY OUTCOMES:
Pain scores during mobilisation 24h | 24 hours after end of surgery
  Pain scores (visual analogue scale (VAS 0-100 mm; no pain = 0; worst imaginable pain = 100)) with active 30 degrees flexion of the hip
Pain scores at rest 24h | 24 hours after end of surgery
  Pain scores at rest (VAS 0-100 mm; no pain = 0; worst imaginable pain = 100)
Maximum level of pain | 24 hours after end of surgery
  Maximum level of pain (VAS 0-100 mm No pain = 0; worst imaginable pain = 100) during walk of 5 meters
Adverse events in the intervention period | From end of surgery + 24 hours
  Proportion of patients with one or more AEs in the intervention period

OTHER OUTCOMES:
Serious adverse events within one year | Within 90 days
  SAEs, including death, within 90 days after surgery defined as SAE (according to ICH-GCP-guidelines) except 'prolongation of hospitalisation' that has been modified to 'prolongation of hospitalization with ≥4 days'
Pain scores during mobilisation 6h | 6 hours after end of surgery
  Pain scores (visual analogue scale (VAS 0-100 mm; no pain = 0; worst imaginable pain = 100)) with active 30 degrees flexion of the hip
Pain scores at rest 6h | 6 hours after end of surgery
  Pain scores at rest (VAS 0-100 mm; no pain = 0; worst imaginable pain = 100)
Prevalence of nausea | 6 and 24 hours after end of surgery
  Prevalence of nausea, 6 and 24 hours after end of surgery
Number of vomiting episodes | 0-24 after end of surgery. Reported by interview 24 hours after end of surgery
  The number of productive vomiting events (volume estimated over 10 ml) is recorded corresponding to the period 0-24 hours
Consumption of ondansetron and dehydrobenzperidole | 0-24 hours after end of surgery
  Consumption of ondansetron and dehydrobenzperidole in mg
Incidence of dizziness during 5 meter walk | 24 hours after end of surgery
  Incidence of dizziness during 5 meter walk 24 hours after surgery
Blood loss | Intraoperatively
  Blood loss in ml during the surgical procedure
Quality of sleep | 24 hours after end of surgery
  Quality of sleep (VAS 0-100 mm; worst possible sleep = 0; best possible sleep = 100) Worst possible sleep = 0; best possible sleep = 100
Days alive and outside hospital within 90 days after surgery | Within 90 days after surgery
  Days alive and outside hospital within 90 days after surgery
Oxford Hip Score at 90 days | At 90 days after surgery
  5-point Lipert-scale (no, mild, moderate, severe and extreme)
Quality of life (EQ-5D-5L) at 90 days | At 90 days after surgery
  EuroQol five-dimensions 5 point Lipert scale (EQ-5D-5L)
Opioid use at 90 days | Within 90 days after surgery
  Consumption of opioids within 90 days after surgery
Serious adverse events within 1 year | Within one year after surgery
  Proportion of participants with one or more serious adverse events, including death, within one year after surgery, according to ICH-GCP guidelines[24] (except for 'prolongation of hospitalization' that has been modified to 'prolongation of hospitalization with ≥4 days')
Oxford Hip Score at one year | One year after surgery
  5-point Lipert-scale (no, mild, moderate, severe and extreme)
Quality of life (EQ-5D-5L) at one year | One year after surgery
  EuroQol five-dimensions 5 point Lipert scale (EQ-5D-5L)
Opioid use at one year | Within one year after surgery
  Consumption of opioids within one year after surgery

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (7):
  - Næstved-Slagelse-Ringsted Hospitals, Næstved, Danmark
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Hellerup
  - Hillerød Hospital, Hillerød
  - Køge Hospital, Køge
  - Odense University Hospital (OUH), Odense
  - Svendborg Hospital, Svendborg

REFERENCES:
- [Derived] Steiness J, Hagi-Pedersen D, Lunn TH, Overgaard S, Brorson S, Graungaard BK, Lindberg-Larsen M, Varnum C, Lundstrom LH, Beck T, Skettrup M, Pedersen NA, Bieder MJ, von Cappeln AG, Pleckaitiene L, Lindholm P, Bukhari SSH, Derby CB, Nielsen MG, Exsteen OW, Vinstrup LO, Thybo KH, Gasbjerg KS, Norskov AK, Jakobsen JC, Mathiesen O; RECIPE trial group. Non-opioid analgesic combinations following total hip arthroplasty (RECIPE): a randomised, placebo-controlled, blinded, multicentre trial. Lancet Rheumatol. 2024 Apr;6(4):e205-e215. doi: 10.1016/S2665-9913(24)00020-1. Epub 2024 Mar 5. PMID 38458208
- [Derived] Steiness J, Hagi-Pedersen D, Lunn TH, Lindberg-Larsen M, Graungaard BK, Lundstrom LH, Lindholm P, Brorson S, Bieder MJ, Beck T, Skettrup M, von Cappeln AG, Thybo KH, Gasbjerg KS, Overgaard S, Jakobsen JC, Mathiesen O. Paracetamol, ibuprofen and dexamethasone for pain treatment after total hip arthroplasty: protocol for the randomised, placebo-controlled, parallel 4-group, blinded, multicentre RECIPE trial. BMJ Open. 2022 Sep 1;12(9):e058965. doi: 10.1136/bmjopen-2021-058965. PMID 36190737
- See also: Trial website — http://www.recipetrial.com